CLINICAL TRIAL: NCT04898725
Title: Effects of Vitamin D Supplementation on Depression and Inflammatory Markers in Adolescent and Youth With Major Depression and Vitamin D-deficiency: a Partially Randomized Preference Trial in Taiwan
Brief Title: Effects of Vitamin D Supplementation on Depression and Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shen-Ing,Liu, Senior Attending Psychiatrist, Professor, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 109-2314-B-195 -017 -MY3
Record Dates: First submitted 2021-05-04; First posted 2021-05-24 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Major Depression; Vitamin D Deficiency
MeSH Terms: conditions — Depressive Disorder, Major; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vit D Group (randomized) (Experimental): Subjects will be randomly assigned to receive a daily vitamin D supplementation (4800IU daily) for 8 weeks
  Interventions: Dietary Supplement: Vitamin D3
- Control Group (randomized) (No Intervention): Subjects will be randomly assigned to receive a placebo for 8 weeks.
- Preference Vit D Group (non-randomized) (Experimental): Subjects with a strong preference to receive a daily vitamin D supplementation (4800IU daily) for 8 weeks.
  Interventions: Dietary Supplement: Vitamin D3
- Preference no Vit D Group (non-randomized) (No Intervention): Subjects with a strong preference to receive usual care (not receiving vitamin D supplements) for 8 weeks.

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 4800IU daily
  Arms: Preference Vit D Group (non-randomized); Vit D Group (randomized)

SUMMARY:
The current study is designed as a prospective partially randomized patient preference (PRPP) trial and recruit psychiatric outpatients or inpatients. Participants who agree to receive randomization will be randomly assigned into a supplementation or placebo group, after stratification for pre-intervention vitamin D status (12-20 ng/mL or <12 ng/mL) and depression status (HDRS-17 ≥ 17 or < 17). Participants who decline randomization but agree to receive follow-up in the observational cohort choose their preferred method (either 4800 IU vitamin D3 per day, or usual care without supplementation). Severity of depression, any change of medication, and side effect will be assessed at baseline and at 2-week intervals for 8 weeks. Serum levels of 25(OH)D, C-Reactive protein (CRP) and 12 cytokines, anthropometrical measurements, dietary intake, physical activity and sun exposure will be assessed at baseline and post-intervention. Additionally, serum levels of 25(OH)D will be assessed at 4 weeks to ensure its safety level.

DETAILED DESCRIPTION:
Investigators will conduct a partially randomized patient preference (PRPP) trial and recruit psychiatric outpatients or inpatients. Inclusion criteria are young people aged 10 to 24, fulfilling the DSM-V criteria of major depressive disorder (MDD) with scores of HDRS-17≥10, psychotropic medication have been kept unchanged for a month and will remain unchanged during intervention period, and serum 25-hydroxycholecalciferol (25-OH-D) levels lower than 20 ng/ml. Exclusion criteria are comorbid with organic mental disorders, alcohol or substance use disorders, schizophrenia, delusion disorder, bipolar disorder, autistic spectrum disorder, anorexia nervosa, and IQ less than 70; endocrine disorders including diabetes, thyroid and parathyroid disorder; serious neurological disorders including epilepsy, severe traumatic brain injury, and neurodegenerative conditions; liver disease, kidney disease, heart disease or other serious health conditions; use drug interfering with vitamin D metabolism.

Participants who agree to receive randomization will be randomly assigned into a supplementation or placebo group, after stratification for pre-intervention vitamin D status (12-20 ng/mL or <12 ng/mL) and depression status (HDRS-17 ≥ 17 or < 17). Supplementation arm will receive oral dose 4800 IU vitamin D3 per day (three soft capsules of 800 IU vitamin D, twice a day) and placebo arm will receive placebo every day (three soft capsules with identical appearance, twice a day) for 8 weeks. Both groups continue to receive standard psychiatric care by child psychiatrists. Randomization and allocation will be concealed from researchers, participants and treating physicians. Participants who decline randomization but agree to receive follow-up in the observational cohort choose their preferred method (either 4800 IU vitamin D3 per day, or usual care without supplementation). Severity of depression, any change of medication, and side effect will be assessed at baseline and at 2-week intervals for 8 weeks. Serum levels of 25(OH)D, CRP and 12 cytokines, anthropometrical measurements, dietary intake, physical activity and sun exposure will be assessed at baseline and post-intervention. Additionally, serum levels of 25(OH)D will be assessed at 4 weeks to ensure its safety level.

ELIGIBILITY:
Inclusion Criteria:

* 1.patients who attend psychiatric outpatient clinics or who are admitted to the psychiatric inpatient ward at the above sites.
* 2.clinical diagnosis of depression-related disorders and scores of HDRS-17 ≥ 10.
* 3.psychotropics have been kept unchanged for at least a month.
* 4.aged 10 to 24.
* 5.serum 25-hydroxycholecalciferol (25-OH-D) levels lower than 20 ng/ml.

Exclusion Criteria:

* 1.endocrine disorders

  1. including diabetes
  2. thyroid
  3. parathyroid disorder.
* 2.serious neurological disorders

  1. epilepsy
  2. severe traumatic brain injury
  3. neurodegenerative conditions
* 3.liver disease
* 4.kidney disease
* 5.heart disease
* 6.other serious health conditions.
* 7.severe mental disorders

  1. Organic mental disorders
  2. Alcohol or substance use disorders active within 3 months
  3. Schizophrenia
  4. Delusional disorder
  5. Psychotic disorders not elsewhere classified.
  6. Bipolar disorder.
  7. Autistic spectrum disorder.
  8. Anorexia nervosa.
  9. Mental retardation with IQ less than 70.
  10. High violence or suicide risk.
* 8.Patients use drugs or herbals interfering with vitamin D metabolisms

  1. phenobarbital
  2. phenytoin
  3. anti-tuberculosis drugs
  4. thiazide diuretics.
* 9.Pregnant or expect to be pregnant during study participation.

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 142 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change of total score of 17-item Hamilton Depression Rating Scale (HDRS-17) | baseline and at 8 weeks (the end of intervention)
  17-item Hamilton Depression Rating Scale is an interview-based instrument for rating the overall levels of severity of the symptoms of depression and the response to treatment. Each item is rated from 0 to 4 or 0 to 2; the scores correspond to increases in severity. Total scores range from 0 to 52.

SECONDARY OUTCOMES:
17-item Hamilton Depression Rating Scale (HDRS-17) | change from baseline score at 8 weeks
  HDRS-17 is measured totally 5 times, at week 0, 2 weeks, 4 weeks, 6 weeks, 8 weeks. The change in total HDRS-17 score between baseline and the intermediate 2-week, 4-week, 6-week follow-ups were considered secondary outcomes measures.
Response rate of 17-item Hamilton Depression Rating Scale (HDRS-17) | at 2 weeks, 4 weeks, 6 weeks, 8 weeks
  Response rate is defined as a reduction in HDRS-17 total score of at least 50 percent relative to the beginning of the randomized phase (baseline).
Remission rate of 17-item Hamilton Depression Rating Scale (HDRS-17) | at week 2, 4, 6, 8 weeks
  Remission rate is defined as an absolute HDRS-17 total score of ≤ 7 at each follow-up assessment.
End of intervention remission rate in17-item Hamilton Depression Rating Scale (HDRS-17) | at 8 weeks
  Remission rate is defined as an absolute HDRS-17 total score of ≤ 7 at the end of treatment (8 week after intervention).
Change of total score of Beck Depression Inventory-Second Edition | change from baseline score at 8 weeks
  Beck Depression Inventory is a 21-item self-report measure, scored from 0 to 3 (range 0-63), and greater scores indicate severe depression symptoms.Beck Depression Inventory (BDI) is measured totally 5 times, at week 0, 2 weeks, 4 weeks, 6 weeks, 8 weeks. The change in total BDI score between baseline and each of follow-ups (2-week, 4-week, 6-week, 8-week follow-ups) were considered secondary outcomes measures.
Significant change (mean±SD) in vitamin D status | baseline and at 8 weeks
  serum levels of 25(OH)D, units of measure is ng/mL

OTHER OUTCOMES:
Change of total score of Generalized Anxiety Disorder Questionnaire | baseline and at 8 weeks (the end of intervention)
  Generalized Anxiety Disorder Questionnaire is a 7-item self-report measure, scored from 0 to 3 (range 0-21), and greater scores indicate severe anxiety symptoms.
Significant change (mean±SD) in serum concentration of hs-CRP | baseline and 8 weeks after intervention
  The serum concentration of hs-CRP (mg/L) will be measured at baseline and 8 weeks after intervention. Normal range is <0.3 mg/L.
Significant change (mean±SD) in serum concentration of cytokine targets | baseline and 8 weeks after intervention
  The serum concentration of cytokine targets (IL-1β, IL-2, IL-6, IL-12, IL-15, TNF-α, IFN-γ, IL-4, IL-5, IL-13, IL-10, IL-1Ra) (unit: pg/mL) will be measured at baseline and 8 weeks after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Shen-Ing Liu, PhD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No